CLINICAL TRIAL: NCT06172231
Title: Effects of Instrument Assisted Soft Tissue Mobilization in Addition to Conventional Physiotherapy in Knee Arthrofibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2023/25
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Knee Arthrofibrosis
Keywords: Knee, Arthrofibrosis,IASTM Instrument Assisted Soft Tissue Mobilization,range of motion

STUDY DESIGN:
Intervention Model Description: Both group will be recruited concurrently. Both group will receive treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A ( Conventional physiotherapy) (Active Comparator): 5 min moist Hot pack ,Patellar joint mobilizations and Tibiofemoral ,Maitland grades III and IV (5 oscillations in first week) ,PROMs of knee joint ( 5 reps) ,Quad sets ( 5 reps with 5 sec hold)Progression: 5 repetition of each exercise would be add in every week ,Frequency: 4 sessions in 4-week period Duration: 15_ 35 min each session.
  Interventions: Procedure: Conventional therapy
- Group B ( IASTM along with conventional physiotherapy)) (Experimental): rst conventional Physiotherapy same as group A thenIASTM protocol.The treatment processes consist of Four phases: warm up (heat), Graston Technique®, passive stretching and cryotherapy.6_10 long strokes on Hamstring and Rectus femoris by using G1 instrument .Brief bouts (30 - 60 s) of deeper and more specific.Frequency: 4 sessions in 4-week period.Duration: 15_35 min each session.
  Interventions: Procedure: Instrument Assisted Soft tissue mobilization; Procedure: Conventional therapy

INTERVENTIONS:
Procedure: Instrument Assisted Soft tissue mobilization — The treatment processes consist of Four phases: warm up (heat), Graston Technique®, passive stretching and cryotherapy.6_10 long strokes on Hamstring and Rectus femoris by using G1 instrument .Brief bouts (30 - 60 s) of deeper and more specific. Frequency: 4 sessions in 4-week period. Duration: 15_35 min each session.
  Arms: Group B ( IASTM along with conventional physiotherapy))
Procedure: Conventional therapy — 5 min moist Hot pack ,Patellar joint mobilizations and Tibiofemoral ,Maitland grades III and IV (5 oscillations in first week) ,PROMs of knee joint ( 5 reps) ,Quad sets ( 5 reps with 5 sec hold)Progression: 5 repetition of each exercise would be add in every week ,Frequency: 4 sessions in 4-week period Duration: 15_ 35 min each session.

SUMMARY:
Arthrofibrosis is the abnormal proliferation of fibrous tissue within a joint and around the joint that leads to loss of motion, pain, muscle weakness, swelling, functional limitation. Study conducted to determine additional effects of IASTM along with conventional physiotherapy as compared to conventional physiotherapy alone on Range of motion, functional limitation and pain in knee arthrofibrosis.

DETAILED DESCRIPTION:
Arthrofibrosis is common condition after surgeries, most of the arthrofibrosis literature addresses arthrofibrosis after arthroplasty or ligamentous reconstruction, and it is replete with manipulation under anesthesia or with arthroscopic interventions or both. Study will be conducted over period of 1 year at fauji foundation hospital.Ethical approval from ERC foundation university medical college. Participants recruited and written inform consent, following which they will be required to complete a self-reported demographic form. The data will be entered and analyzed on SPSS 22. IASTM is simple and effective intervention to improve Rom and functional limitation in patients with knee arthrofibrosis

ELIGIBILITY:
Inclusion Criteria:

* post Total knee replacement patients
* Extension lag >10
* Flexion deficit >25
* Age 18_60
* both male and female
* Numeric pain rating scale between 3-5

Exclusion Criteria:

* skin allergy
* Diabetic patient
* Any vascular disease
* Prolonged use of Corticosteroids
* Any infective or active inflammatory condition
* Fracture or dislocation
* Lower extremity functional scale score above 71.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Lower Extremity Functional Scale | 4 weeks
  The Lower Extremity Functional Scale (LEFS), developed by the North American Orthopaedic Rehabilitation Research Network, consists of 20 items. Each item is scored from 0 (extreme difficulty/unable to perform activity) to 4 (no difficulty), for a total maximum score of 80 points, which indicates a high functional level. The LEFS scores demonstrated excellent test-retest reliability (intraclass correlation coefficients ranging between 0.85 and 0.99
Knee range of motion | 4 weeks
  Goniometer use to check range of motion of knee joint.For range of motion, intertester reliability (r = .98; ICC = .99) and validity (r = .97-.98; ICC = .98-.99)
pain intensity | 4 weeks
  The Numeric pain rating scale is an 11 point scale comprising a number from 0 through 10, 0 indicates no pain and 10 indicates worst imaginable pain

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan